CLINICAL TRIAL: NCT07311226
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of IBI3033 in Healthy Participants
Brief Title: A First-in-human, Single-ascending-dose Study of IBI3033 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI3033A101
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- IBI3033 Dose 1 subcutaneously (SC) (Experimental)
  Interventions: Drug: IBI3033
- Placebo IV (Placebo Comparator)
  Interventions: Drug: Placebo
- IBI3033 Dose 3 SC (Experimental)
  Interventions: Drug: IBI3033
- IBI3033 Dose 2 intravenously (IV) (Experimental)
  Interventions: Drug: IBI3033
- IBI3033 Dose 2 SC (Experimental)
  Interventions: Drug: IBI3033
- Placebo SC (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Participants in placebo group will receive placebo SC/IV.
  Arms: Placebo IV; Placebo SC
Drug: IBI3033 — Participants in IBI3033 group will receive a signle dose of IBI3033 at the protocol specified dose SC/IV.
  Arms: IBI3033 Dose 1 subcutaneously (SC); IBI3033 Dose 2 SC; IBI3033 Dose 2 intravenously (IV); IBI3033 Dose 3 SC

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of IBI3033 in Chinese healthy participants. The entire trial cycle includes a 4-week screening period, 1-day treatment period and 12-week follow-up period.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males/females aged 18-55 years (inclusive).
2. BMI 18.0-28.0 kg/m²; weight ≥50 kg (male) or ≥45 kg (female).
3. Willing to use effective contraception for 6 months post-dosing.

Exclusion criteria:

1. History of blood or needle sickness, or those who cannot tolerate venipuncture.
2. Female participants who are pregnant or breastfeeding at screening or randomization.
3. History of severe infection or significant injury within 6 months, or surgery within 3 months, or any infection requiring systemic medication within 1 month prior to screening.
4. History of live or attenuated vaccination within 1 month prior to screening, or those who plan to be vaccinated during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs)/serious adverse events (SAEs) | Baseline to Day 85
  Percentage of participants who have experienced AEs/SAEs

SECONDARY OUTCOMES:
PK parameter: Cmax | Baseline to Day 85
  Observed maximum plasma concentration of IBI3033
PK parameter: tmax | Baseline to Day 85
  Time to achieve Cmax of IBI3033
PK parameter: AUC | Baseline to Day 85
  Area under the plasma concentration-time curve of IBI3033
Immunogenticity profiles | Baseline to Day 85
  Frequency of anti-drug antibody (ADA) of IBI3033

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China